CLINICAL TRIAL: NCT04970303
Title: The Roles of Endocrine Disrupting Chemicals, Growth Hormone and Thyroid Function in Attention-deficit/Hyperactivity Disorder
Brief Title: Endocrine Disrupting Chemicals and Hormones in ADHD
Acronym: ADHD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Liang-Jen, Professor and Visiting Staff, Chang Gung Memorial Hospital
Other Study IDs: 201900376A3
Record Dates: First submitted 2021-07-01; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; endocrine disrupting chemicals; growth hormone; thyroid; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Thyroid Diseases | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: investigator will recruit 60 patients with ADHD (aged between 6 and 16). Blood (10 ml) and urine (10 ml) will be obtained from each participant to analyze the levels of EDCs (Phthalates, Phenols and Parabens), growth hormone and thyroid function (TSH, T3, Free T4, T4, growth hormone, IGF-1and IGF-BP3). Behavior symptoms (ADHD-RS and SNAP-IV) and neuropsychological function (WISC, CPT and CATA) of each participant will be assessed. Patients with ADHD will receive treatment in a clinical practice and then will be followed up for 12 months. At the 12th month, the same procedures as those performed at the baseline will be replicated for patients with ADHD.
  Interventions: Drug: Methylphenidate
- Control group: investigator will recruit 60 age- and gender-matched control subjects. Blood (10 ml) and urine (10 ml) will be obtained from each participant to analyze the levels of EDCs (Phthalates, Phenols and Parabens), growth hormone and thyroid function (TSH, T3, Free T4, T4, growth hormone, IGF-1and IGF-BP3). Behavior symptoms (ADHD-RS and SNAP-IV) and neuropsychological function (WISC, CPT and CATA) of each participant will be assessed.

INTERVENTIONS:
Drug: Methylphenidate — Retina or Concerta
  Other Names: used Retina or Concerta
  Groups: Case group

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a common neurodevelopmental disorder in children and adolescents. Growth hormone and thyroid function are associated with both physical and neurocognitive development. Endocrine disrupting chemicals (EDCs) could disturb the normal function of endocrine systems, and further link to the pathophysiology of ADHD. In addition, whether methylphenidate for treating ADHD influences growth hormone and thyroid function of patients remains unclear.

DETAILED DESCRIPTION:
Therefore, this study aims (1) to investigate the prospective role of EDCs, growth hormone and thyroid function in clinical manifestations of ADHD; and (2) to determine the influence of pharmacotherapy on growth hormone and thyroid function among patients with ADHD under a one-year methylphenidate treatment.

Methods: In this two-year study, we will recruit 120 patients with ADHD (aged between 6 and 16) and 120 age- and gender-matched control subjects. Blood (10 ml) and urine (10 ml) will be obtained from each participant to analyze the levels of EDCs (Phthalates, Phenols and Parabens), growth hormone and thyroid function (TSH, T3, Free T4, T4, growth hormone, IGF-1and IGF-BP3). Behavior symptoms (ADHD-RS and SNAP-IV) and neuropsychological function (WISC, CPT and CATA) of each participant will be assessed. Patients with ADHD will receive treatment in a clinical practice and then will be followed up for 12 months. At the 12th month, the same procedures as those performed at the baseline will be replicated for patients with ADHD.

This study will provide proof of the relationships of EDCs, endocrine systems and ADHD manifestations in clinical samples and further explain the biological pathogenesis of ADHD. In addition, this study will elucidate the influence of ADHD medications on growth hormone and thyroid function. Such information may become an important reference for future research and safety of pharmacotherapy for patients with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADHD aged between 6 and 16.
* The patients were either newly diagnosed with ADHD or had an existing diagnosis but had not taken medication for ADHD during the previous 6 months or more.

Exclusion Criteria:

* Patients with a history of major physical or additional psychiatric diseases

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 patients with ADHD (aged between 6 and 16) and 60 age- and gender-matched control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth hormone and thyroid function | Baseline
  IGF-1 (ng/mL), insulin-like growth factor-1; IGFBP-3 (ng/mL), IGF binding protein-3; TSH (µIU/mL), thyroid-stimulating hormone; T3 (ng/dL), triiodothyronine; T4 (µg/dL), thyroxine
Growth hormone and thyroid function | month 12
  IGF-1 (ng/mL), insulin-like growth factor-1; IGFBP-3 (ng/mL), IGF binding protein-3; TSH (µIU/mL), thyroid-stimulating hormone; T3 (ng/dL), triiodothyronine; T4 (µg/dL), thyroxine

SECONDARY OUTCOMES:
Children's growth-Height | Baseline
  Height (cm)
Children's growth-Height | month 12
  Height (cm)
Children's growth-body weight | Baseline
  body weight (kg)
Children's growth-body weight | month 12
  body weight (kg)

OTHER OUTCOMES:
ADHD clinical symptoms, The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | Baseline
  The SNAP-IV is a 26-item questionnaire used to evaluate ADHD symptoms and severity that needs to be completed by parents or teachers. The 26 items include 18 for ADHD symptoms (nine for inattention and nine for hyperactivity/impulsivity) and eight for oppositional defiant disorder (ODD) symptoms as defined by the DSM-IV. Each item is scored from 0-3 on a Likert scale. The total scores are ranged between 0 (min) to 78 (max), and higher scores mean a greater severity of ADHD.
ADHD clinical symptoms, The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | month 12
  The SNAP-IV is a 26-item questionnaire used to evaluate ADHD symptoms and severity that needs to be completed by parents or teachers. The 26 items include 18 for ADHD symptoms (nine for inattention and nine for hyperactivity/impulsivity) and eight for oppositional defiant disorder (ODD) symptoms as defined by the DSM-IV. Each item is scored from 0-3 on a Likert scale. The total scores are ranged between 0 (min) to 78 (max), and higher scores mean a greater severity of ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, MD, MPH, PhD, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Liang-Jen Wang, Kaohsiung City, Taiwan